CLINICAL TRIAL: NCT03992846
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Study to Assess the Efficacy and Safety of Linzagolix in Subjects With Moderate to Severe Endometriosis-associated Pain.
Brief Title: Efficacy and Safety of Linzagolix for the Treatment of Endometriosis-associated Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-OBE2109-003
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2022-06

CONDITIONS: Endometriosis
Keywords: Dysmenorrhea; Dyspareunia; Dyschezia; Non-menstrual pelvic pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Dyspareunia; Constipation | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Linzagolix 75 mg (Experimental)
  Interventions: Drug: 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule
- Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg) (Experimental)
  Interventions: Drug: 200 mg linzagolix tablet; Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg); Drug: Placebo tablet to match 75 mg linzagolix tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo tablet to match 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule

INTERVENTIONS:
Drug: 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg) — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg); Placebo
Drug: Placebo tablet to match 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg; Placebo
Drug: Placebo capsule to match Add-back capsule — For oral administration once daily
  Arms: Linzagolix 75 mg; Placebo

SUMMARY:
The primary objective of this study is to demonstrate the efficacy and safety of linzagolix administered orally once daily for 3 months at a dose of 75 mg alone or of 200 mg in combination with add-back hormone replacement therapy (ABT: estradiol (E2) 1 mg / norethisterone acetate (NETA) 0.5 mg) versus placebo, in the management of moderate to severe endometriosis-associated pain (EAP).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study to demonstrate the efficacy and safety of linzagolix administered orally once daily at doses of 75 mg alone and 200 mg in combination with low dose ABT (E2 1 mg/NETA 0.5 mg) versus placebo in the management of moderate to severe EAP in 450 women.

Eligible subjects who have completed the 6-month treatment period may enter a separate extension study for 6 additional months of active treatment (no placebo control). Subjects who do not continue in the extension study will enter a 6 month treatment-free follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

The subject must have:

* Her most recent surgical and - if available - histological diagnosis of pelvic endometriosis up to 10 years before screening.
* Moderate to severe endometriosis-associated pain during the screening period.
* Regular menstrual cycles.
* BMI ≥ 18 kg/m2 at the screening visit. -

Exclusion Criteria:

The subject will be excluded if she:

* Is pregnant or breast feeding or is planning a pregnancy within the duration of the treatment period of the study.
* Is less than 6 months postpartum or 3 months postabortion/ miscarriage at the time of entry into the screening period.
* Has had a surgical history of any major abdominal surgery within 6 months or any interventional surgery for endometriosis performed within a period of 2 months before screening.
* Did not respond to prior treatment with GnRH agonists or GnRH antagonists for endometriosis.
* Has a history of, or known, osteoporosis or other metabolic bone disease.
* Has chronic pelvic pain that is not caused by endometriosis and requires chronic analgesic or other chronic therapy which would interfere with the assessment of endometriosis-associated pain.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females Only
Enrollment: 486 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecomte, Study Director — ObsEva SA
Locations (71):
- United States (22):
  - Achieve Clinical Research/ ID # 601, Birmingham, Alabama
  - Choice Research, LLC/ ID # 609, Dothan, Alabama
  - Southeast Clinical Research/ ID # 618, Chiefland, Florida
  - Universal Axon - Homestead, LLC/ ID # 620, Homestead, Florida
  - Multi-Specialty Research Associates, Inc./ ID # 625, Lake City, Florida
  - Wellington Anti-Aging, LLC/ ID # 613, Loxahatchee Groves, Florida
  - Adventura Clinical Research/ ID # 616, Miramar, Florida
  - Stedman Clinical Trials/ ID # 612, Tampa, Florida
  - Advanced Specialty Research/ ID # 610, Nampa, Idaho
  - Affinity Clinical Research Institute/ ID # 622, Oak Brook, Illinois
  - Women's & Family Care, LLC dba GTC Research/ ID # 608, Shawnee Mission, Kansas
  - Southern Clinical Research / ID # 611, Metairie, Louisiana
  - Quad Clinical Research LLC/ ID # 615, St Louis, Missouri
  - The Center for Women's Health & Wellnes/ ID # 603, Lawrenceville, New Jersey
  - PMG Research of Wilmington/ ID # 614, Wilmington, North Carolina
  - UWCR - Lyndhurst Clinical Researc/ ID# 605, Winston-Salem, North Carolina
  - Obstetrics & Gynecology Associates, Inc./ ID# 606, Fairfield, Ohio
  - Invocare Medical Research & Healthcare Center/ ID # 607, West Columbia, South Carolina
  - Chattanooga Medical Research LLC/ ID# 602, Chattanooga, Tennessee
  - Next Innovative Clinical Research/ ID # 617, Houston, Texas
  - Storks Research, LLC/ ID # 623, Sugar Land, Texas
  - Tanner Clinic/ ID # 624, Layton, Utah
- Austria (3):
  - Salzburger Landeskliniken / ID # 105, Salzburg
  - AKH Vienna University of Medicine Vienna / ID # 101, Vienna
  - AKH Vienna University of Medicine Vienna/ ID # 103, Vienna
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Sliven/ ID # 131, Sliven
  - MHAT Dr. Bratan Shukerov / ID #138, Smolyan
  - Medical Centre Excelsior /ID # 135, Sofia
  - Group Practice for Specialized Medical Assistance in GINART/ ID # 132, Sofia
  - Multiprofile Hospital for Active Treatment St. Sofia/ ID # 137, Sofia
  - University Multiprofile Hospital for Active Treatment "Sofiamed"/ ID # 133, Sofia
- Czechia (3):
  - MUDr Jan Drahonovsky, Ustav pro peci o matku a dite/ ID #163, Prague
  - Gynekologicko - Porodnicka Ambulance/ ID # 162, Tábor
  - Gynekologie MU Dr.Lubomir Mikulasek / ID # 160, Újezd nad Lesy
- France (3):
  - CHRU Besançon Hopital/ ID # 204, Besançon
  - CHRU Strasbourg - Hopital Hautepierre/ ID # 205, Strasbourg
  - Clinique Pasteur / ID # 206, Toulouse
- Hungary (4):
  - Principal SMO Kft/ ID # 250, Baja, Bács-Kiskun county
  - Róbert Károly Magánkórház/ ID # 253, Budapest
  - Szent Anna Szuleszeti-Nogyogyaszati/ ID # 251, Debrecen
  - Mediroyal Prevencios Kozpont/ ID # 252, Kecskemét
- Poland (11):
  - Lubelskie Centrum Diagnostyczne/ ID # 402, Świdnik, Lublin Voivodeship
  - Prywatna Klinika Ginekologiczno - Położnicza/ ID # 404, Bialystok, Podlaskie Voivodeship
  - VITA LONGA Sp. z o.o./ ID # 408, Katowice
  - Clinical Medical Research sp. Z o. O/ ID # 406, Katowice
  - Indywidualna Specjalistyczna Praktyka Lekarska Krzysztof Wilk/ ID # 411, Katowice
  - Niepubliczny Zaklad Opieki Zrowotnej GynCentrum/ ID # 407, Katowice
  - Kotarski Jan Specjalistyczny Gabinet Ginekologiczno Polozniczy/ ID # 405, Lublin
  - Centrum Medyczne Chodźki Lublin/ ID # 403, Lublin
  - Centrum Ginekologii Endokrynologii i Medycyny Rozrodu "Artemida"/ ID # 409, Olsztyn
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu/ ID # 410, Przemyśl
  - Specjalistyczny Gabinet Lekarski Krzysztof Dynowski / ID # 401, Warsaw
- Romania (6):
  - Quantum Medical Center SRL/ ID # 353, Bucharest
  - Centrul Medical EUROMED/ ID # 351, Bucharest
  - Spitalul Clinic "Nicolae Malaxa"/ ID # 352, Bucharest
  - Sp Cl de Obstetrica si Ginecologie "Prof. Dr. Panait Sirbu"/ ID # 354, Bucharest
  - Gine Plus SRL Cluj- Napoca/ ID # 357, Cluj-Napoca
  - Centrul Medical GALENUS/ ID # 355, Târgu Mureş
- Spain (2):
  - Hospital Regional Universitario de Málaga/ ID # 303, Málaga
  - Hospital General Universitario Reina Sofia/ ID # 304, Murcia
- Ukraine (11):
  - City clinical maternity hospital №1/ ID # 502, Chernivtsi
  - Ivano-Frankivsk regional perinatal center, Family planning center/ ID # 506, Ivano-Frankivsk
  - Kyiv City Maternity Hospital #6/ ID # 504, Kyiv
  - Medical center of LLC "Medical Center "Verum"/ ID # 503, Kyiv
  - Institute of Pediatrics Obstetrics and Gynecology/ ID # 508, Kyiv
  - Kyiv City Clinical Hospital #9/ ID # 501, Kyiv
  - Kyiv City Center of Reproductive and Perinatal Medicine/ ID # 509, Kyiv
  - Ternopil' Communal City Hospital #2/ ID # 511, Ternopil
  - Vinnytsia City Clinical Hospital "Center of Mother and the Child "/ ID # 510, Vinnytsia
  - Zaporizhzhya Regional Clinical Hospital/ ID # 505, Zaporizhzhya
  - Maternity Hospital № 3/ ID # 507, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donnez J, Becker C, Taylor H, Carmona Herrera F, Donnez O, Horne A, Paszkowski M, Petraglia F, Renner SP, Patel A, Boolell M, Bestel E, Dolmans MM. Linzagolix therapy versus a placebo in patients with endometriosis-associated pain: a prospective, randomized, double-blind, Phase 3 study (EDELWEISS 3). Hum Reprod. 2024 Jun 3;39(6):1208-1221. doi: 10.1093/humrep/deae076. PMID 38648863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 854 subjects screened, 486 were randomized. Between randomization and Day 1 (i.e., first day of dosing), 2 subjects in the LGX 75 mg group discontinued due to protocol deviation. Thus, 484 randomized subjects were treated and comprised the FAS and SAF.
Pre-assignment Details: Participants with a diagnosis of endometriosis were enrolled in a 1:1:1 ratio in one of three treatment groups: Linzagolix (=LGX) 75 mg, LGX 200 mg+Add-back (=ABT) or Placebo.
Groups:
- LGX 75 mg: One Linzagolix 75 mg tablet, One Linzagolix 200 mg matching placebo tablet and one Add-back matching placebo capsule were administered once daily orally for 6 months.
- LGX 200 mg+ABT: One Linzagolix 200 mg tablet, One Linzagolix 75 mg matching placebo tablet and one Add-back capsule (E2 1 mg / NETA 0.5 mg) were administered once daily orally for 6 months.
- Placebo: One Linzagolix 75 mg matching placebo tablet, one Linzagolix 200 mg matching placebo tablet and one Add-back matching placebo capsule were administered once daily orally for 6 months.
Period: Overall Study
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Started | 160 | 162 | 162
Month 3 | 149 | 155 | 149
Month 6 | 140 | 143 | 137
Completed | 140 | 143 | 137
Not Completed | 20 | 19 | 25
Not completed — Adverse Event | 8 | 6 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Pregnancy | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal by Subject | 8 | 10 | 20
Not completed — Sponsor decided to exclude the patient | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo | Total
Number analyzed (Participants) | 160 | 162 | 162 | 484
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 160 | 162 | 162 | 484
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (6.4) | 34.6 (6.8) | 34.9 (6.8) | 34.9 (6.6)
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 35.5 [31.0 to 40.0] | 35.0 [30.0 to 40.0] | 35.0 [31.0 to 40.0] | 35.0 [30.0 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 162 | 162 | 484
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 1 | 13
  Not Hispanic or Latino | 155 | 155 | 161 | 471
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 158 | 159 | 160 | 477
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 0 | 0 | 1 | 1
  Romania | 18 | 12 | 19 | 49
  Hungary | 0 | 0 | 2 | 2
  United States | 7 | 12 | 7 | 26
  Czechia | 2 | 3 | 1 | 6
  Ukraine | 70 | 63 | 70 | 203
  Poland | 58 | 64 | 57 | 179
  Bulgaria | 4 | 5 | 4 | 13
  France | 0 | 1 | 0 | 1
  Spain | 1 | 2 | 1 | 4
Weight [Mean (Standard Deviation); unit: kg] | 67.73 (14.45) | 65.75 (14.75) | 65.81 (11.96) | 66.42 (13.77)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.60 (5.23) | 24.09 (5.17) | 24.14 (4.44) | 24.27 (4.95)

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Dysmenorrhea (DYS) at Month 3 - Proportion of Responders
Description: Percentage of subjects with reduction of 1.1 for DYS in mean pelvic pain score within last 28 days prior to Month 3 or discontinuation, and stable or decreased use of analgesics for Endometriosis-associated pain (=EAP) within the same calendar days.
Time Frame: Baseline to Month 3
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Number analyzed (Participants) | 160 | 162 | 162
Percentage of responders | 44.0 [36.3 to 52.0] | 72.9 [65.3 to 79.4] | 23.5 [17.5 to 30.7]
Statistical Analysis 1: Comparison: LGX 75 mg vs Placebo; Test type: Other — The criterion for defining a subject as a responder over the last 28 days of randomized treatment up to Month 3 was a reduction of 1.10 or greater from baseline pain for Dysmenorrhea (DYS); p < 0.001, Bonferroni-corrected p-value; Odds Ratio (OR) = 2.56, 97.5% CI 2-sided [1.46 to 4.49]
Statistical Analysis 2: Comparison: LGX 200 mg+ABT vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bonferroni-corrected p-value; Odds Ratio (OR) = 8.80, 97.5% CI 2-sided [4.86 to 15.91]

2. Primary Outcome: Reduction of Non-menstrual Pelvic Pain (NMPP) at Month 3 - Proportion of Responders
Description: Percentage of subjects with reduction of 0.8 for NMPP in mean pelvic pain score within last 28 days prior to Month 3 or discontinuation, and stable or decreased use of analgesics for Endometriosis-associated pain (=EAP) within the same calendar days.
Time Frame: Baseline to Month 3
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
Number analyzed (Participants) | 160 | 162 | 162
Percentage of responders | 38.9 [31.5 to 46.9] | 47.3 [39.5 to 55.3] | 30.9 [24.1 to 38.6]
Statistical Analysis 1: Comparison: LGX 75 mg vs Placebo; Test type: Other — The criterion for defining a subject as a responder over the last 28 days of randomized treatment up to Month 3 was a reduction of 0.80 or greater from baseline pain for Non-Menstrual Pelvic Pain (NMPP); p = 0.279, Bonferroni-corrected p-value; Odds Ratio (OR) = 1.43, 97.5% CI 2-sided [0.83 to 2.45]
Statistical Analysis 2: Comparison: LGX 200 mg+ABT vs Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.007, Bonferroni-corrected p-value; Odds Ratio (OR) = 2.01, 97.5% CI 2-sided [1.18 to 3.42]

ADVERSE EVENTS:
Time Frame: Day 1 to Month 6 of the treatment period
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial subject administered an investigational medicinal product (IMP) and which did not necessarily have a causal relationship with this treatment. Therefore, AE was any unfavorable sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/162 | 0/162
Serious Adverse Events (participants affected / at risk) | 1/160 | 2/162 | 0/162
Other Adverse Events (participants affected / at risk) | 83/160 | 94/162 | 69/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=160) | LGX 200 mg+ABT (N=162) | Placebo (N=162)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=160) | LGX 200 mg+ABT (N=162) | Placebo (N=162)
Hot flush (Vascular disorders) | 12 (15) | 11 (11) | 4 (4)
Headache (Nervous system disorders) | 13 (17) | 17 (24) | 13 (25)
Fatigue (General disorders) | 6 (6) | 11 (11) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 10 (13)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (5) | 6 (7) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 5 (5)
Mood swings (Psychiatric disorders) | 8 (8) | 5 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 2 (2)
COVID-19 (Infections and infestations) | 5 (5) | 6 (6) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03992846/Prot_002.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03992846/SAP_003.pdf